CLINICAL TRIAL: NCT07131410
Title: Efficacy of Hyaluronic Acid Cream in Preventing Foot Ulceration Risk in Patients With Type 2 Diabetes and Moderate-to-Severe Peripheral Neuropathy
Brief Title: Efficacy of Hyaluronic Acid Cream in Preventing Foot Ulceration Risk in Patients With Type 2 Diabetes and Moderate-to-Severe Peripheral Neuropathy: A Randomized Clinical Trial.
Acronym: HIALU_PREV_FOO
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaga (Other)
Responsible Party: Principal Investigator, Gabriel Gijon-Nogueron, Efficacy of Hyaluronic Acid Cream in Preventing Foot Ulceration Risk in Patients with Type 2 Diabetes and Moderate-to-Severe Peripheral Neuropathy: A Randomized Clinical Trial., University of Malaga
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: Universidad Miguel Hernández
Record Dates: First submitted 2024-11-09; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: DIABETES
Keywords: WOUND; DIABETIC FOOT
MeSH Terms: conditions — Diabetes Mellitus; Wounds and Injuries; Diabetic Foot

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients who apply 10% urea daily (Sham Comparator): Participants will apply a 10% urea cream following the same protocol. Patients will receive the container cream for application on both feet after thoroughly washing and drying them. It is recommended to use an amount the size of a hazelnut for each foot, spreading it in a thin layer over the entire foot, excluding the interdigital area. The application will be done every night for twelve months. The product will be massaged into the foot for 15 seconds. During the study, participants will not be allowed to use any other topical product (cream, emulsion, gel, lotion, or oil) on their feet and/or nails.
  Interventions: Other: Group hialuronyc
- Patients who apply hyaluronic acid daily (Experimental): Patients will receive the container with Hialucic® cream for application on both feet after thoroughly washing and drying them. It is recommended to use an amount the size of a hazelnut for each foot, spreading it in a thin layer over the entire foot, excluding the interdigital area. The application will be done every night for twelve months. The product will be massaged into the foot for 15 seconds. During the study, participants will not be allowed to use any other topical product (cream, emulsion, gel, lotion, or oil) on their feet and/or nails.
  Interventions: Other: Group hialuronyc

INTERVENTIONS:
Other: Group hialuronyc — Patients will receive the container with cream for application on both feet after thoroughly washing and drying them. It is recommended to use an amount the size of a hazelnut for each foot, spreading it in a thin layer over the entire foot, excluding the interdigital area. The application will be done every night for twelve months. The product will be massaged into the foot for 15 seconds. During the study, participants will not be allowed to use any other topical product (cream, emulsion, gel, lotion, or oil) on their feet and/or nails.

SUMMARY:
A triple-blind randomized clinical trial aimed at evaluating the efficacy of a hyaluronic acid cream in preventing foot ulcers in patients with type 2 diabetes and moderate-to-severe peripheral neuropathy.

The primary objective is to determine the effectiveness of this cream in preventing ulcerations after 12 months of use in this population, compared to the use of another cream containing 10% urea. Secondary objectives include assessing changes in hydration, skin stiffness, and pH across various areas of the foot, with results compared between the intervention and control groups.

The study will be conducted at Miguel Hernández University between 2025 and 2027. A total of 166 adult participants with type 2 diabetes and moderate-to-severe peripheral neuropathy will be randomized into two groups: the intervention group, which will apply the hyaluronic acid cream daily, and the control group, which will use a 10% urea cream. Measurements of skin hydration, pH, and stiffness, along with the xerosis index, will be taken during three scheduled visits (at 3, 6, and 12 months). Neuropathy will be assessed through sensitivity and reflex tests, while sociodemographic and clinical variables will be recorded at the start of the study.

Participants will log their treatment adherence and any potential adverse effects through a mobile application. The data obtained on skin hydration, pH, and stiffness will be analyzed to identify differences between the two groups, with differences considered statistically significant if p < 0.05.

This study aims to provide evidence on the effectiveness of hyaluronic acid in preventing ulcerations and improving skin characteristics of the foot in patients with diabetes and peripheral neuropathy.

DETAILED DESCRIPTION:
Hypothesis

The hypothesis is that the daily application of a cream with hyaluronic acid on the foot does not reduce the incidence of foot ulcers in patients with type 2 diabetes and moderate-to-severe peripheral neuropathy after one year of follow-up, compared to the application of a cream with 10% urea.

Primary Objective

Evaluate the efficacy of topical hyaluronic acid cream over 12 months in preventing foot ulceration in patients with moderate-to-severe peripheral neuropathy, compared to the application of a cream with 10% urea.

Secondary Objectives

Determine the average hydration level of different foot areas (forefoot, midfoot, and hindfoot) in patients with diabetes and peripheral neuropathy.

Assess the degree of stiffness in different foot areas (forefoot, midfoot, and hindfoot) in patients with diabetes and peripheral neuropathy.

Measure the skin pH of various foot regions (forefoot, midfoot, and hindfoot) in patients with diabetes and peripheral neuropathy.

Compare the hydration, stiffness, and pH results between the intervention and control groups after applying hyaluronic acid cream on the foot for 12 months.

Methodology

This is a triple-blind, randomized clinical trial in which patient assignment will be performed using a random number table, managed by the researcher responsible for each patient. Sampling will be consecutive and carried out at the podiatry clinic of Miguel Hernández University between 2025 and 2027.

Each patient will be randomly assigned to a group:

Group A (Intervention Group): Patients will apply a hyaluronic acid cream daily to both feet for 12 months.

Group B (Control Group): Patients will apply a 10% urea cream following the same protocol as Group A.

The study will be conducted in accordance with the principles of the Declaration of Helsinki and submitted for approval by the relevant Ethics Committee. Written informed consent will be obtained from each patient before any procedures are conducted.

Participants will be recruited from San Juan Health Center and the Endocrinology Service of San Juan de Alicante Hospital, with five physicians and ten nurses from both centers involved in recruitment.

Inclusion Criteria

Adults aged 18 or older, diagnosed with type 2 diabetes and moderate-to-severe peripheral neuropathy (diagnosed with a score ≥6 on the Michigan scale), who have not used any topical moisturizer or keratolytic agents on their feet for at least two weeks prior.

Exclusion Criteria

Presence of ulcerative skin lesions on the foot Diagnosed peripheral arterial disease, indicated by the absence of both peripheral pulses and/or Ankle-Brachial Index less than 1 or greater than 1.4 Dermatological diseases affecting foot hydration: atopic dermatitis, ichthyosis, or psoriasis Use of custom-made plantar orthoses, as the material could affect foot hydration Sample Size Calculation Assuming an annual ulceration incidence of 20% in patients with moderate-to-severe peripheral neuropathy and expecting an incidence of 5% in the treated group, the required sample size is 83 subjects per group (75 + 10% for attrition), with a 95% confidence level (alpha risk 5%) and an 80% statistical power (beta risk 20%).

Clinical Interview

During a clinical interview, sociodemographic variables such as gender and age will be collected. For diabetes mellitus (DM), the number of years since diagnosis, usual control parameters, and current pharmacological treatment will be documented. Smoking status will be classified as non-smoker, former smoker, or current smoker, including time smoked or time since quitting. Weekly physical activity will also be recorded.

Examination

Patient weight (kg) and height (cm) will be measured using a Bamed® scale with a stadiometer to calculate body mass index (BMI) according to the formula: weight (kg)/height² (m). Subjects will be classified based on WHO criteria into normal weight (BMI 18.50-24.99), overweight (BMI 25-29.9), and obesity (BMI ≥30).

Blood pressure (systolic and diastolic in mmHg) will be measured using an Omron® automatic sphygmomanometer.

Metabolic control will be assessed via a blood test conducted within six months prior to inclusion. Quantitative variables to be recorded include: total cholesterol (mg/dL), LDL cholesterol (mg/dL), HDL cholesterol (mg/dL), triglycerides (mg/dL), fasting blood glucose (mg/dL), HbA1c (%), estimated glomerular filtration rate (eGFR) in mL/min/1.73 m², and urine albumin-to-creatinine ratio.

Peripheral Neuropathy Assessment

Peripheral neuropathy will be evaluated using the Michigan Neuropathy Screening Instrument (MNSI), involving a brief physical examination that includes:

Foot inspection for deformities, dry skin, hair or nail abnormalities, calluses, or infections.

Vibration sensation on the dorsal surface of the big toe assessed with a 128Hz Rydel-Seiffer tuning fork, with three measurements considered abnormal if the average score is ≤6 for patients under 60 and ≤4 for those over 80.

Achilles reflex assessment: Using a reflex hammer on the Achilles tendon; plantar flexion is rated as present. Reflexes requiring the Jendrassik maneuver are marked as "present with reinforcement," and reflexes that remain absent are considered absent.

Pressure sensation with the monofilament at 10 anatomical points on the foot. Skin Assessment

The following measurements will be performed at eight foot locations (pulp of the first, third, and fifth toes, metatarsal heads of the first, third, and fifth metatarsals, and medial and lateral plantar surfaces of the heel):

Hydration: Using the Corneometer CM 825, which measures stratum corneum hydration.

Skin pH: Measured with a glass electrode on the skin surface. Stiffness: Using the Indentomer IDM 800 to assess skin rigidity. Cream Treatment Evaluation

Adverse Effects: Local adverse signs and symptoms, including pruritus, erythema, stinging, and dermal lesions, will be recorded in each visit using a mobile app designed for this purpose.

Adherence: Participants will use a project-specific app to log their adherence to the treatment.

Pre-ulcerous or Ulcerous Lesions: The presence of dermal lesions will be recorded, detailing their location, type, and size. Participants may communicate any dermal lesions to the investigator through the app and will be evaluated at the university clinic outside of study follow-up visits.

Methodology

The cream will be packaged in two opaque containers labeled A and B, with no indication of their contents. Neither the patient nor the researcher will know the contents of each container or the patient's assigned group. Both groups will follow the same application instructions.

Group A (Intervention Group): Participants will apply the Hialucic® cream to both feet nightly for twelve months.

Group B (Control Group): Participants will apply a 10% urea cream following the same protocol.

Assessment Schedule

At the start of the study (D0) At 3 months (M3) At 6 months (M6) At 12 months (M12)

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 or older, diagnosed with type 2 diabetes and moderate-to-severe peripheral neuropathy (diagnosed with a score ≥6 on the Michigan scale), who have not used any topical moisturizer or keratolytic agents on their feet for at least two weeks prior

Exclusion Criteria:

* Presence of ulcerative skin lesions on the foot Diagnosed peripheral arterial disease, indicated by the absence of both peripheral pulses and/or Ankle-Brachial Index less than 1 or greater than 1.4 Dermatological diseases affecting foot hydration: atopic dermatitis, ichthyosis, or psoriasis Use of custom-made plantar orthoses, as the material could affect foot hydration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2026-11-15 (Estimated); Study Completion 2027-03-15 (Estimated)

PRIMARY OUTCOMES:
Photo analysis | 12 months
  The occurrence of dermal lesions on the skin will be recorded, specifying their location, type, and size. The patient will be able to report any dermal lesion to the investigator via the app, and the lesion will be assessed at the university clinic, regardless of the study's scheduled follow-up visit

CONTACTS AND LOCATIONS:
Locations (1):
- University of Malaga, Málaga, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fitzner A, Knuhr K, Brandt M, Bielfeldt S. Investigating the effect of the pH of foot care product formulations on pedal skin in diabetic and non-diabetic subjects. Int J Cosmet Sci. 2023 Aug;45(4):524-538. doi: 10.1111/ics.12861. Epub 2023 Apr 27. PMID 37014141
- [Result] Garrigue E, Martini J, Cousty-Pech F, Rouquier A, Degouy A. Evaluation of the moisturizer Pedimed((R)) in the foot care of diabetic patients. Diabetes Metab. 2011 Sep;37(4):330-5. doi: 10.1016/j.diabet.2010.12.004. Epub 2011 Feb 23. PMID 21349756
- [Result] Federici A, Federici G, Milani M. An urea, arginine and carnosine based cream (Ureadin Rx Db ISDIN) shows greater efficacy in the treatment of severe xerosis of the feet in Type 2 diabetic patients in comparison with glycerol-based emollient cream. A randomized, assessor-blinded, controlled trial. BMC Dermatol. 2012 Sep 25;12:16. doi: 10.1186/1471-5945-12-16. PMID 23009311
- [Result] Cristaudo A, Francesconi L, Ambrifi M, Frasca M, Cavallotti C, Sperduti E. Efficacy of an emollient dermoprotective cream in the treatment of elderly skin affected by xerosis. G Ital Dermatol Venereol. 2015 Jun;150(3):297-302. PMID 25946673
- [Result] Couteau C, Coiffard LJ, Sebille-Rivain V. Influence of excipients on moisturizing effect of urea. Drug Dev Ind Pharm. 2006 Feb;32(2):239-42. doi: 10.1080/03639040500466361. PMID 16537204
- [Result] Chicharro-Luna E, Zunica-Garcia S, Martinez-Algarra C, Gracia-Sanchez A. Age-related variations in stratum corneum hydration in the foot. Maturitas. 2024 Nov;189:108104. doi: 10.1016/j.maturitas.2024.108104. Epub 2024 Aug 22. PMID 39180901